CLINICAL TRIAL: NCT02938715
Title: Pilot Study of the Pragmatic Use of Mobile Phone Based Follow up of Actinic Keratoses Treated With Topical 5-fluorouracil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 955458
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

ARMS (2):
- Feedback group (teledermatology) (Experimental)
  Interventions: Other: teledermatology feedback
- Control group (phone only) (No Intervention)

INTERVENTIONS:
Other: teledermatology feedback — subject provided feedback to continue or discontinue their cream (based on actinic keratoses grading and lesion counting)
  Arms: Feedback group (teledermatology)

SUMMARY:
In this study, subjects who are attending the dermatology clinic and who have already been prescribed topical 5-fluorouracial for the treatment of actinic keratoses as part of their standard of care will be recruited. The purpose of the study is to assess patient satisfaction when engaging in follow up treatment of actinic keratosis via the HIPAA-compliant teledermatology platform called Klara. Additionally, the goal is to assess the difference in total duration of treatment between treatment and control group. A total of 50 subjects will be enrolled and will be randomly assigned into the treatment group (teledermatology group; n=25) or control group (telephone only group; n=25).

DETAILED DESCRIPTION:
Objectives

To assess patient satisfaction when engaging in follow up treatment of actinic keratoses: Follow up of subjects with actinic keratoses (AK) who have been prescribed topical 5-fluorouracil (5-FU) therapy as part of their standard of care.

To assess the difference in total dose of exposure to 5-FU between treatment and control group.

Background

Teledermatology is a growing field within dermatology that has started to adapt the use of mobile phone technology (1). The growth of teledermatology has allowed greater access to care in both the inpatient and outpatient setting (1, 2), as well as in educational services (3). The aim of this study is to investigate how mobile phone photographic teledermatology can be adapted for use in the dermatology clinic to continually engage with the patient. More specifically, the researchers seek to understand how mobile phone technology can be used in the evaluation of subjects on topical 5-FU therapy for their actinic keratoses.

Diffuse actinic damage is typically treated with field therapy (4) that involves the use of topical 5-FU. Patients are advised to apply the cream twice daily for 2-4 weeks (5). However, many patients note misunderstanding with these instructions (6). Typical follow up has included telephone based grading and in person follow up (5). However, a return visit to the clinic can be both burdensome to the patient and fill up the clinic with follow up appointments instead of allowing the appointment slot to go to examination of a new patient, thereby reducing access to care for other patients. Telephone conversations are not based on a physical exam and thus do not allow for objective evaluation of the treatment area. For this reason, the researchers seek to use mobile phone photography to evaluate patients with actinic keratoses on topical 5-FU treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age or older
* Subjects who have already been prescribed topical 5-fluorouracil for treatment of scalp, facial, arm, or hand actinic keratoses but have not initiated treatment yet

Exclusion Criteria:

* Adults unable to consent
* Non English speaking or illiterate
* Subjects with known allergy to 5-fluorouracil
* Subjects who do not have access to a smartphone capable of engaging with the online teledermatology platform
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Difference in total dose of exposure to 5-FU between teledermatology and control group (measured as days of exposure x frequency of application per day) | 4 weeks
  The total exposure to 5-FU will be calculated as total doses over 4 week period.

SECONDARY OUTCOMES:
Patient satisfaction assessment | 4 weeks and 8 weeks
Change in clinical grading of actinic keratoses | baseline and weeks 1, 2, 3, 4, 8
Change in AK lesion count | baseline and weeks 1, 2, 3, 4, 8
Change in severity of symptoms | baseline and weeks 1, 2, 3, 4, 8
Difference in adverse effects including erythema, pruritus, burning, soreness, and/or tenderness, crusting and/or erosions, scaling and/or flaking, and swelling | baseline and weeks 1, 2, 3, 4, 8
Difference in number of clinic visits between the 2 groups | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Department of Dermatology, Sacramento, California, United States

REFERENCES:
- [Background] Zuo KJ, Guo D, Rao J. Mobile teledermatology: a promising future in clinical practice. J Cutan Med Surg. 2013 Nov-Dec;17(6):387-91. doi: 10.2310/7750.2013.13030. PMID 24138974
- [Background] Fox LP. Practice Gaps. Improving accessibility to inpatient dermatology through teledermatology. JAMA Dermatol. 2014 Apr;150(4):424-5. doi: 10.1001/jamadermatol.2013.9516. No abstract available. PMID 24522259
- [Background] Brewer AC, Endly DC, Henley J, Amir M, Sampson BP, Moreau JF, Dellavalle RP. Mobile applications in dermatology. JAMA Dermatol. 2013 Nov;149(11):1300-4. doi: 10.1001/jamadermatol.2013.5517. PMID 24067948
- [Background] Stockfleth E, Peris K, Guillen C, Cerio R, Basset-Seguin N, Foley P, Sanches J, Culshaw A, Erntoft S, Lebwohl M. A consensus approach to improving patient adherence and persistence with topical treatment for actinic keratosis. Int J Dermatol. 2015;54(5):509-15. doi: 10.1111/ijd.12840. Epub 2015 Apr 10. PMID 25865875
- [Background] Pomerantz H, Hogan D, Eilers D, Swetter SM, Chen SC, Jacob SE, Warshaw EM, Stricklin G, Dellavalle RP, Sidhu-Malik N, Konnikov N, Werth VP, Keri J, Lew R, Weinstock MA; Veterans Affairs Keratinocyte Carcinoma Chemoprevention (VAKCC) Trial Group. Long-term Efficacy of Topical Fluorouracil Cream, 5%, for Treating Actinic Keratosis: A Randomized Clinical Trial. JAMA Dermatol. 2015 Sep;151(9):952-60. doi: 10.1001/jamadermatol.2015.0502. PMID 25950503
- [Background] Esmann S, Jemec GB. Patients' perceptions of topical treatments of actinic keratosis. J Dermatolog Treat. 2014 Oct;25(5):375-9. doi: 10.3109/09546634.2012.757285. Epub 2013 Feb 24. PMID 23215635